CLINICAL TRIAL: NCT00350701
Title: Effect of Androgel on Inflammatory Mediators and Oxidative Stress in Type 2 Diabetic Males With Hypogonadism
Brief Title: Effect of Androgel on Type 2 Diabetic Males With Hypogonadism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, MD, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1911
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus Type 2
Keywords: DM type 2; Hypogonadism; Testosterone; AndroGel
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- androgel 5g (Experimental): androgel 5g
  Interventions: Drug: androgel
- androgel 10g (Experimental): androgel 10g
  Interventions: Drug: androgel 10g
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: androgel — androgel 5g
  Arms: androgel 5g
Drug: androgel 10g — androgel 10g
  Other Names: androgel
  Arms: androgel 10g
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This is to study the effect of replacing testosterone on different inflammatory cells in type 2 diabetics with low testosterone levels.

DETAILED DESCRIPTION:
Type 2 diabetes is an atherosclerotic, pro-inflammatory and pro-oxidative stress. Hypogonadism( low testosterone) is also associated with increased levels of inflammatory mediators and atherosclerosis.

This project is about studying the effect of testosterone replacement on different inflammatory cells in blood and urine. It will also compare the dose dependent effect on inflammatory cells. This also involves comparing level of inflammation in hypogonadic diabetic males treated with testosterone with those not treated with any replacement therapy.

This study involves applying AndroGel for 8 wks and studying effects during this time and thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Males with age 35-75 years inclusive.
* Evidence of hypogonadism: low free testosterone.
* Type 2 Diabetes
* People on stable doses of cholesterol lowering medications, blood pressure medications and multi-vitamins are allowed.
* If currently on testosterone replacement,testosterone treatment will be held for 8 weeks.
* BP under control even if on medication.

Exclusion Criteria:

* Coronary event or procedure in previous past 4 wks.
* High PSA
* H/O prostate cancer
* Hepatic or renal disease
* Participation in any other concurrent clinical trial
* Any other life- threatening , non cardiac disease.
* Uncontrolled BP
* Congestive heart failure
* High hemoglobin
* Use of investigational agent or therapeutic regimen within 30 days of study.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-07; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — Kaleida Health/Diabetes Endocrinology Center of WNY
Locations (1):
- Diabetes-Endocrinology Center of Western NY, 115 flint road, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Androgel 5g | Androgel 10g | Placebo
Started | 17 | 17 | 15
Completed | 17 | 17 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgel 5g | Androgel 10g | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 15 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 12 | 39
  >=65 years | 4 | 3 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (8) | 57 (9) | 59 (9) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 17 | 17 | 15 | 49

OUTCOME MEASURES:

1. Primary Outcome: Effect of Androgel Treatment on Relative Nuclear Factor kB Activity Compared to Placebo
Description: To measure the percent change from baseline at 8 weeks in Nuclear Factor kB DNA binding activity (in arbitrary units normalized to 100% at baseline) between AndroGel and Placebo using electrophoretic mobility shift assay (EMSA). Values at 8 weeks are converted to percent change and compared between the groups
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Androgel 5g | Androgel 10g | Placebo
Number analyzed (Participants) | 17 | 17 | 15
Percent change from baseline
  baseline | 100 (0) | 100 (0) | 100 (0)
  8 week | 236 (197) | 82 (61) | 100 (103)

2. Secondary Outcome: Effect of Androgel Treatment on Reactive Oxygen Species Generation Compared to Placebo
Description: Comparison of relative percent change from baseline at 8 weeks in reactive oxygen species generation (measured as arbitrary units normalized to 100% at baseline) in mononuclear cells after either AndroGel or placebo using chemiluminescence PMSF activation assay. Values at 8 weeks are converted to percentage of the baseline and compared between the groups
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of baseline value
Arm/Group | Androgel 5g | Androgel 10g | Placebo
Number analyzed (Participants) | 17 | 17 | 15
percentage of baseline value
  baseline | 100 (0) | 100 (0) | 100 (0)
  8 week | 91 (8) | 125 (17) | 110 (17)

3. Secondary Outcome: Change in Inflammatory Mediator C-Reactive Protein (CRP) Following Treatment With Testosterone
Description: To measure the relative percent change from baseline in the inflammatory mediator (CRP) at 8 weeks (values in ng/ml normalized to100% at baseline) following treatment with androgel compared to placebo. Values (in ng/ml) are converted to percentage of baseline at 8 weeks.
Time Frame: 8 week
Measure: Mean (Standard Deviation); unit: percentage of baseline value
Arm/Group | Androgel 5g | Androgel 10g | Placebo
Number analyzed (Participants) | 17 | 17 | 15
percentage of baseline value
  baseline | 100 (0) | 100 (0) | 100 (0)
  8 week | 68 (9) | 130 (18) | 95 (10)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Androgel 5g | Androgel 10g | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes